CLINICAL TRIAL: NCT01066169
Title: Immune Response After Vaccination Against Pandemic A/H1N1 Influenza in the Immunocompromised Host. Vaccination Response in ImmunoCompromised Host
Brief Title: Vaccination Response in ImmunoCompromised Host. Immune Response After Vaccination Against Pandemic A/H1N1 Influenza
Acronym: RICH-3
Status: Completed | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: D. Soonawala, MD, Leiden University Medical Center
Other Study IDs: P09.187
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2012-01-30 (Estimated); Status verified 2010-02

CONDITIONS: HIV
Keywords: Pandemic Influenza A/H1N1; HIV; Antibodies; Replicaton
MeSH Terms: interventions — lactitol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, Plasma, Peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy volunteers: Healthy subjects without HIV, vaccinated with Pandemic Influenza A/H1N1
  Interventions: Biological: Foceteria® (Novartis)
- HIV-infected patients: HIV-infected patients, vaccinated with Pandemic Influenza A/H1N1
  Interventions: Biological: Foceteria® (Novartis)

INTERVENTIONS:
Biological: Foceteria® (Novartis) — This is not an interventional study. In this observational study we monitored the immune response in a cohort of people who were vaccinated during the national vaccination campaign. The vaccine that was used in The Netherlands is the monovalent influenza A/California/2009(H1N1) MF59-adjuvanted surface-antigen vaccine. It contains 7,5 µg hemagglutinine and the MF59C.1 adjuvant, which is an oil-in-water emulsion, composed of Squalene 9.75 mg, Polysorbate 80 1.175 mg and Sorbitan trioleate 1.175 mg. This vaccine has been approved for use according to a two dose schedule.

SUMMARY:
As recommended by the Dutch Health Council, certain risk groups and health care workers in The Netherlands were vaccinated to prevent morbidity due to pandemic influenza A/H1N1. Adults were vaccinated twice with the monovalent influenza A/California/2009(H1N1) MF59-adjuvanted surface-antigen vaccine Focetria® (Novartis). The vaccination campaign was executed by general practitioners.

The aim of the study is to verify whether HIV-infected individuals generate an adequate immune response after the first and after the second vaccination.

DETAILED DESCRIPTION:
AIM OF THIS STUDY:

Primary objective: Do HIV-infected individuals mount a protective humoral response following vaccination for pandemic influenza A/H1N1 with the monovalent influenza A/California/2009(H1N1) MF59-adjuvanted surface-antigen vaccine Focetria® (Novartis).

Secondary objective: 1) To evaluate the strength of the immune response in HIV-infected individuals compared to healthy volunteers. 2) To evaluate whether a second dose, administered at least 21 days after the first increases the proportion of HIV-infected individuals that have a titer above the threshold associated with protection. 3) To assess whether vaccination is associated with an increases in HIV-replication. 4) To assess whether very early antibody responses occur, which may may indicate immunological memory, for example due to cross reactivity from past influenza infection or vaccination.

STUDY DESIGN:

This is not an interventional study. In this single-centre observational study we will monitor the immune response in a cohort of people who are to be vaccinated during the national vaccination campaign.

Population: The population base for this study consists of HIV-infected adult outpatients at our hospital and of healthy hospital employees. All Dutch and English speaking HIV-infected LUMC outpatients above 18 years of age, on a stable antiretroviral regimen or not yet in need of treatment, are sent a letter inviting them to take part. Healthy hospital employees are invited to take part with a letter, which is handed out upon vaccination. Inclusion is possible until three days after the first vaccination. Exclusion criteria are: use of systemic immunosuppressive medication, an ongoing infection, recent flu-like symptoms and pregnancy. The following characteristics are documented at baseline: age, gender, co-morbidity, medication, year of prior influenza vaccinations and year of diagnosis of HIV infection. All participants are requested to fill out standardized diary assessing flu-like symptoms and use of new medication during the 60 day follow-up.

Laboratory analysis: Lymphocyte counts are determined at baseline, prior to vaccination. A serum sample is taken prior to the first vaccination (day -30 to day 0), prior to the second vaccination (day 17-20) and after the second vaccination (day 60). Viral load is determined at baseline (day -30 to day 0) and after the second vaccination (day 5-7) in a subgroup of 10 persons with undetectable viral load at the preceding outpatient visit. Antibody responses are detected in duplicate for each sample by means of hemagglutination-inhibition (HI) assays according to standard methods at the Erasmus Medical Center in Rotterdam.

Statistical analysis: No formal sample-size calculation was performed. We intend to include a maximum of 100 subjects with HIV and 50 healthy hospital employees. The crude outcome estimates will be adjusted for variables that may influence the outcome (age, CD4 lymphocyte count, use of HAART, viral load).

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years of age
* Stable antiretroviral regimen or not yet in need of treatment (in case of HIV-infected patients)

Exclusion Criteria:

* Use of systemic immunosuppressive medication
* An ongoing infection
* Recent flu-like symptoms and pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV patients at the department 'Infectious Diseases' of the Leiden University Medical Centre and healthy volunteers (hospital employees of the Leiden University Medical Centre)
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2009-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Antibody titer after second vaccination | day 55-60

SECONDARY OUTCOMES:
Antibody titer after second vaccination | day 17-20
Antibody titer shortly after first vaccination (day 5-7) | day 5-7
HIV replication after vaccination | day 5-7

CONTACTS AND LOCATIONS:
Overall Officials: Frank P Kroon, MD PhD, Principal Investigator — Leiden University Medical Centre; Leo G Visser, MD PhD, Study Chair — Leiden University Medical Centre; Luc BS Gelinck, MD, Study Chair — Leiden University Medical Centre; A F Rimmelzwaan, Prof PhD, Study Chair — Leiden University Medical Centre; Darius Soonawala, MD, Study Director — Leiden University Medical Centre
Locations (1):
- Leiden University Medical Centre, Leiden, South Holland, Netherlands

REFERENCES:
- [Derived] Soonawala D, Rimmelzwaan GF, Gelinck LB, Visser LG, Kroon FP. Response to 2009 pandemic influenza A (H1N1) vaccine in HIV-infected patients and the influence of prior seasonal influenza vaccination. PLoS One. 2011 Jan 31;6(1):e16496. doi: 10.1371/journal.pone.0016496. PMID 21304982
- See also: Publication of results — http://www.plosone.org/article/info%3Adoi%2F10.1371%2Fjournal.pone.0016496